CLINICAL TRIAL: NCT05842018
Title: Toripalimab in Combination With Chemotherapy and Antiangiogenic Agents in Patients With Non Small Cell Lung Cancer After Failure of Immunotherapy (PD-1/L1 Inhibitors): a Prospective, Single-arm, Phase II Trial
Brief Title: Toripalimab in Combination With Chemotherapy and Antiangiogenic Agents in Patients With Non-Small Cell Lung Cancer After Failure of Immunotherapy (PD-1/L1 Inhibitors)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-NSCLC-CO396
Record Dates: First submitted 2023-04-24; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-03

CONDITIONS: Non Small Cell Lung Cancer Recurrent
MeSH Terms: interventions — toripalimab; anlotinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab, Chemotherapy and Antiangiogenic Agents (Experimental)
  Interventions: Drug: Toripalimab, Anlotinib and Chemotherapy

INTERVENTIONS:
Drug: Toripalimab, Anlotinib and Chemotherapy — Combination therapy:
  Toripalimab 240mg will be intravenously administered on Day 1, Q3W; anlotinib: 12 mg qd d1-d14, d15-d21 discontinued, Q3W; investigator selected chemotherapy regimen (paclitaxel, pemetrexed or gemcitabine and other chemotherapeutic drugs which were not administered in the first-line therapy) for a total of 4 cycles.
  Maintenance therapy:
  After combination therapy, Patients who achieved complete response（CR）, partial response (PR), or stable disease (SD) were administered with toripalimab plus anlotinib as maintenance therapy. until disease progression or intolerable toxicity, treatment for 2 years, investigator decision, withdrawal of consent, or death.
  Other Names: JS001

SUMMARY:
This is a phase II, single arm, open-label, single-center study to evaluate the efficacy and safety of Toripalimab combined with Chemotherapy and Antiangiogenic Agents in patients with Non-Small Cell Lung Cancer After Failure of Immunotherapy (PD-1/L1 inhibitors)

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily participate in this study, signed and dated informed consent with good compliance and follow-up;
* Diagnosed as locally advanced and / or metastatic non-small cell lung adenocarcinoma (NSCLC) by cytology or histology;
* First-line PD-1/PD-L1 inhibitors treatment failure;
* Provide detectable specimens (tissue or blood) for genotyping before enrollment, and the patients should be with negative EGFR and ALK gene test results;
* Had at least one measurable lesion according to RECIST 1.1 criteria
* Anticipated overall survival more than 3 months;
* ECOG (Eastern Cooperative Oncology Group) scale 0-2;
* Normal organ function and bone marrow function;
* Resistant to first-line immune checkpoint inhibitor therapy and discontinued for more than 4 weeks;
* Women of childbearing age must have taken reliable contraceptive measures and performed a pregnancy test (serum or urine) within 7 days prior to enrollment, and the results were negative, and were willing to use appropriate methods during the trial and 4 weeks after the last administration of the test drug.

Exclusion Criteria:

* Patients with small cell lung cancer (including small cell carcinoma and non-small cell carcinoma mixed lung cancer) ;
* Patients who have previously permanently discontinued immunotherapy due to immune-related serious adverse reactions;
* Patients who previously treated with antiangiogenic agents;
* A history of other malignancies within 5 years prior to inclusion, except for cervical carcinoma in situ, basal or squamous cell skin cancer, localized prostate cancer treated with radical surgery, and ductal carcinoma in situ treated with radical surgery;
* Active, known or suspected autoimmune disease;
* Active or chronic hepatitis C or/and hepatitis B infection;
* History of interstitial lung disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Progress free survival | until Progressive Disease (PD) or death (up to 24 months)
  Progress free survival is defined as the time from first dose of study treatment until the first date of either disease progression or death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate | each 21 days up to intolerance the toxicity or PD (up to 24 months)
  Objective response rate is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.prior to progression or any further therapy.
Overall Survival | from first dose of study treatment until death (up to 24 months)
  Overall survival is defined as the time until death due to any cause.
Disease Control Rate | each 21 days up to intolerance the toxicity or PD (up to 24 months)
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.

IPD SHARING:
Plan to Share IPD: No